CLINICAL TRIAL: NCT04635306
Title: Determination of the Effect of 13C-Spirulina Nitrogen Content on In-vivo 13C-Spirulina Gastric Emptying Breath Test (GEBT) Results
Brief Title: 13C-Spirulina Nitrogen Content GEBT Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial results showed no equivalence between GEBT test meals with low nitrogen versus a standard GEBT test meal
Sponsor: Cairn Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-CD-041
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis
Keywords: Gastroenterology; Gastric emptying breath test
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Low Nitrogen GEBT test meal (Experimental): GEBT test meal containing low %N content (below 7%)
  Interventions: Diagnostic Test: Approved GEBT test meal

INTERVENTIONS:
Diagnostic Test: Approved GEBT test meal — FDA-approve GEBT test meal

SUMMARY:
The purpose of this study is to determine whether there is a difference in the human in vivo response to 13C-Spirulina meals manufactured using 13C-Spirulina containing different levels of protein (as measured by %nitrogen).

DETAILED DESCRIPTION:
In this study participants will be administered the standard FDA-approved GEBT in which the test meals contain 13C-Spirulina that has 7.9% Nitrogen content. On a second occasion, a low nitrogen GEBT in which the test meal will contain 13C-Spirulina with a 6.4% Nitrogen content will be administered. Both sets of GEBTs have been manufactured under full cGMPs and both will be administered to the participants according to the FDA-approved GEBT labeling. The two in vivo results of the two independent GEBT test administrations in the study cohort will be compared to determine whether there is any significant different in in vivo 13CO2 signaling.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-85 years old at time of signing consent form
* Ability to eat test meal and provide breath samples

Exclusion Criteria:

* History or physical exam suggestive of systemic disease such as diabetes mellitus or pathophysiologic disorders such as renal failure, chronic heart disease, chronic respiratory disease, liver disease or malabsorption syndrome
* Symptoms consistent with delayed gastric emptying
* History of abdominal surgery except appendectomy
* Use of any medications that may alter gastric motility within two days of the study
* Use of narcotics or anticholinergics within two days of the study
* Females on hormone replacement therapy other than birth control medications
* Receipt of an investigational drug within 4 weeks of the study
* Pregnancy
* Intolerance or allergy to any component of Gastric Emptying Breath Test meal
* History of neurologic or psychiatric disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Difference in vivo 13C-Spirulina GEBT response | Up to 2 weeks
  Determining the difference between measure gastric emptying rate (kPCD) results produced from the low %N 13C-Spirulina GEBT test meal and the FDA-approved test meal

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ryder, MD, PhD, Principal Investigator — Cairn Diagnostics
Locations (1):
- Cairn Diagnostics, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT04635306/Prot_SAP_000.pdf